CLINICAL TRIAL: NCT00123110
Title: Insulin Resistance and Testosterone in Non-Diabetic Postmenopausal Women
Brief Title: Insulin Resistance and Testosterone in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The John A. Hartford Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pennsylvania Diabetes and Endocrinology Research Center (DERC) (Other); TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0031; K23AG019161 (NIH); K23AG1916101A1 (Other Grant/Funding Number: NIA); 5P30DK019525 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Insulin Resistance; Postmenopause
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): metformin pill plus placebo injection
  Interventions: Drug: metformin; Drug: placebo injection
- 2 (Experimental): leuprolide injection plus placebo pill
  Interventions: Drug: leuprolide injection; Drug: placebo pill
- 3 (Placebo Comparator): placebo pill plus placebo injection
  Interventions: Drug: placebo pill; Drug: placebo injection

INTERVENTIONS:
Drug: metformin — Initiated on 500 mg daily and titrated up to 1000 mg twice a day during the first four weeks, remaining at that dose until 12 weeks
  Other Names: Glucophage
  Arms: 1
Drug: leuprolide injection — 3.75 mg injection every 4 weeks (e.g. at baseline, 4, and 8 weeks)
  Other Names: Lupron
  Arms: 2
Drug: placebo pill — matching pill twice a day for 12 weeks
  Arms: 2; 3
Drug: placebo injection — matching injection every 4 weeks (e.g. baseline, 4, and 8 weeks)
  Arms: 1; 3

SUMMARY:
The purpose of this research study is to determine if a relationship between insulin resistance (IR) and testosterone (T) exists in women who have already gone through menopause.

DETAILED DESCRIPTION:
This study tests the central hypothesis that insulin resistance (IR) increases androgen (male sex hormone) production in postmenopausal women. Participation will include five visits, each lasting on average 2.5 hours, over a period of 13-20 weeks.

At the screening visit, the participant's medical history, current use of medications and dietary supplements, and social habits will be recorded. This information will be reviewed on each subsequent visit; participants are asked to maintain their current diet and physical activity level throughout the study.

A brief physical exam will be performed, and blood will be drawn.

At the 2nd (baseline) visit, patients will undergo a euglycemic-hyperinsulinemic clamp (a procedure to measure insulin sensitivity by continuous intravenous infusion of insulin, and variable infusion of glucose). Blood samples will be drawn throughout the procedure. At completion, the insulin infusion will be stopped, participants will be fed, and the glucose infusion continued for at least 15 minutes to ensure stability of the blood glucose concentration. After the procedure, participants will be randomized to receive either metformin plus leuprolide placebo, leuprolide plus metformin placebo, or metformin placebo plus leuprolide placebo. The leuprolide or leuprolide placebo will be administered as an injection by a nurse. The metformin or metformin placebo will be dispensed to the participant in the form of pills, with instructions for titrating the dose. Participants will be contacted by telephone once weekly during the titration period to assess drug tolerability and adverse events (AEs). Participants will be maintained at their maximum tolerated dose for the duration of the study intervention period.

Participants will return every 4 weeks for follow-up. Blood will be drawn, the nurse will administer the leuprolide or leuprolide placebo injection, and metformin or metformin placebo will be dispensed. At the final visit (week 12), participants will undergo a brief physical exam, and will then undergo a final euglycemic-hyperinsulinemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50-79 years with absence of menses for 12 months; for women 50-54 years, Follicle stimulating hormone>30 U/mL to confirm postmenopausal status
* At least one intact ovary
* Free testosterone and fasting insulin levels within required study parameters
* Willing to comply with all study-related procedures
* Capable of giving informed consent

Exclusion Criteria:

* History of cancer requiring treatment within the past 5 years (exceptions may be made by investigator)
* Hospitalization for treatment of vascular disease in the past 6 months
* Uncontrolled hypertension
* Hospitalization for chronic obstructive pulmonary disease or asthma in the past 3 months
* Use of continuous oxygen at home
* Surgery in the last 30 days
* Positive for HIV
* Abnormal blood tests (hemoglobin, fasting triglycerides, fasting glucose, creatinine, liver function)
* History of diabetes mellitus or use of any anti-hyperglycemic medication in the past 3 months
* Disease associated with disordered glucose metabolism (Cushing's disease, acromegaly, pheochromocytoma not surgically cured, chronic pancreatitis)
* History of chronic renal insufficiency
* Intravenous (IV) contrast studies with iodinated materials planned for the 12 week intervention period that cannot be postponed according to the participant's primary care provider
* Acute or chronic metabolic acidosis
* History of liver disease
* Congestive heart failure
* History of androgen-secreting tumors
* Hormone replacement therapy or antiandrogen use in past 6 months
* Use of dehydroepiandosterone (DHEA) or other androgen-containing products in past 6 months
* Corticosteroid use, other than topical, ophthalmic, intraarticular, and inhaled preparations, in past 3 months
* Undiagnosed current vaginal bleeding
* Excessive alcohol intake, either acute or chronic; current illicit substance abuse
* Participation in an investigational drug study within 6 weeks prior to screening visit
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R. Cappola, MD, ScM, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Clinical and Translational Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford ES, Giles WH, Dietz WH. Prevalence of the metabolic syndrome among US adults: findings from the third National Health and Nutrition Examination Survey. JAMA. 2002 Jan 16;287(3):356-9. doi: 10.1001/jama.287.3.356. PMID 11790215
- [Background] Golden SH, Ding J, Szklo M, Schmidt MI, Duncan BB, Dobs A. Glucose and insulin components of the metabolic syndrome are associated with hyperandrogenism in postmenopausal women: the atherosclerosis risk in communities study. Am J Epidemiol. 2004 Sep 15;160(6):540-8. doi: 10.1093/aje/kwh250. PMID 15353414
- [Background] Larsson H, Ahren B. Androgen activity as a risk factor for impaired glucose tolerance in postmenopausal women. Diabetes Care. 1996 Dec;19(12):1399-403. doi: 10.2337/diacare.19.12.1399. PMID 8941471
- [Background] Oh JY, Barrett-Connor E, Wedick NM, Wingard DL; Rancho Bernardo Study. Endogenous sex hormones and the development of type 2 diabetes in older men and women: the Rancho Bernardo study. Diabetes Care. 2002 Jan;25(1):55-60. doi: 10.2337/diacare.25.1.55. PMID 11772901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited beginning 8/11/05 and continued until the last patient was consented on 4/8/08.
Groups:
- Metformin: metformin plus leuprolide placebo (LP) injection
- Leuprolide: leuprolide plus metformin placebo (MP) pill
- Placebo: MP placebo pill plus LP placebo injection
Period: Overall Study
Arm/Group | Metformin | Leuprolide | Placebo
Started | 12 | 12 | 11
Completed | 12 | 12 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Leuprolide | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4) | 58 (7) | 62 (7) | 58 (7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 12 | 12 | 11 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Free Testosterone (T)
Description: Percent change in free T by equilibrium dialysis between baseline and 12 weeks
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Metformin: Randomized to metformin plus leuprolide placebo, treating insulin resistance
- Leuprolide: Randomized to leuprolide plus metformin placebo, pharmacologic lowering of testosterone
- Placebo: Placebo metformin plus placebo leuprolide
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | -6.9 (22.8) | -35.8 (31.8) | 12.1 (17.8)

2. Primary Outcome: Change in Insulin Sensitivity
Description: Change in insulin sensitivity (mg/kg/min) calculated from hyperinsulinemic euglycemic clamp
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
mg/kg/min | 0.44 (0.80) | 0.04 (0.81) | -0.08 (0.73)

3. Secondary Outcome: Percent Change in Luteinizing Hormone (LH) From Baseline
Time Frame: baseline and 12 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | 4.6 [-5.6 to 9.8] | -96.5 [-210.2 to -46.3] | -1.2 [-3.9 to 6.6]

4. Secondary Outcome: Percent Change in Homeostasis Model Assessment Index of Insulin Resistance (HOMA-IR)
Description: Insulin resistance calculated from homeostasis model assessment of insulin resistance (HOMA-IR) equation: fasting insulin x fasting glucose / 405. Higher values indicate more insulin resistance.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | -31.0 (24.39) | -8.18 (35.3) | 4.67 (38.16)

5. Secondary Outcome: Percent Change in Low Density Lipoprotein (LDL)
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | -10.8 (22.2) | 5.3 (19.3) | 25.3 (50.8)

6. Secondary Outcome: Percent Change in Systolic Blood Pressure
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | -4.2 (8.6) | 4.0 (13.6) | -0.3 (8.6)

7. Secondary Outcome: Free T and IR in Women in Whom Metabolic Syndrome is Present vs. Absent
Time Frame: baseline and 12 weeks
Population: Data were not collected and the outcome will never be analyzed.
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Dehydroepiandrosterone Sulfate (DHEA-S)
Time Frame: baseline and 12 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | 2.6 [-10.5 to 18.4] | 0.9 [-15.5 to 21.1] | -2.9 [-17.2 to 8.8]

9. Secondary Outcome: Body Mass Index (BMI)
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin | Leuprolide | Placebo
Number analyzed (Participants) | 12 | 12 | 11
percent change | -1.3 (3.2) | 0.1 (1.5) | 0.3 (1.1)

ADVERSE EVENTS:
Arm/Group | Metformin | Leuprolide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No